CLINICAL TRIAL: NCT02246127
Title: Randomized Open Label Study to Compare the Efficacy and Safety of Everolimus Followed by Chemotherapy With Streptozotocin- Fluorouracilo (STZ-5FU) Upon Progression or the Reverse Sequence, in Advanced Progressive Pancreatic NETs (pNETs)
Brief Title: Sequentiality of Everolimus and STZ-5FU in Advanced Pancreatic Neuroendocrine Tumor
Acronym: SEQTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: European Neuroendocrine Tumor Society (Unknown); Kantar Health (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GETNE1206; 2013-000726-66 (EudraCT Number)
Record Dates: First submitted 2014-08-20; First posted 2014-09-22 (Estimated); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
Keywords: advanced pNET; everolimus; STZ-5FU; treatment sequence
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A, drug: everolimus first (Active Comparator): Everolimus (10mg/daily, oral) followed by STZ-5FU (injection/infusion; Moertel or Uppsala regime).
  Interventions: Drug: Drug: Everolimus; Drug: STZ-5FU
- Sequence B, drug: STZ - 5FU first (Experimental): STZ-5FU (injection/infusion; Moertel or Uppsala regime) followed by Everolimus (10 mg/ daily, oral)
  Interventions: Drug: Drug: Everolimus; Drug: STZ-5FU

INTERVENTIONS:
Drug: Drug: Everolimus — 10mg/daily, oral. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Afinitor
Drug: STZ-5FU — 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-5 every 6 weeks (Moertel) or 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-3, and then 1 day with 1g/m2 and 1 day 400mg/m2 5-FU every 3 weeks (Uppsala).
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: STZ based Chemotherapy

SUMMARY:
The purpose of this study is to compare streptozotocin (STZ) vs everolimus as first line treatment for advanced pNET and to elucidate which sequence of STZ based chemotherapy and the mammalian Target of Rapamycin (mTOR) inhibitor, everolimus, gives better results in terms of second Progression Free Survival (PFS) in well differentiated and advanced pancreatic NETs.

DETAILED DESCRIPTION:
STZ plus 5-Fuorouracil (5FU) is the actual standard of care for advanced pancreatic Neuroendocrine tumours (pNETS) in the European Union. Everolimus has been recently approved for its use in advanced pNETs by the Food and Drug Administration (FDA) and in Europe by the European Medical Agency (EMA).

A randomized study is needed to have a clear knowledge about the best sequence for its administration; this is, before or after palliative chemotherapy.

There may or may not be any benefits from giving first each other treatment of the study. The information obtained from this study will help the physician improve the treatment and management of patients with advanced pNET.

This study was planned to compare STZ-5FU chemotherapy followed by everolimus upon progression versus the reverse sequence. However sequential studies with pNETs are hard to be managed in terms of time and costs. Therefore the protocol was amended to have PFS1 (progression free survival after course 1) as primary endpoint and PFS2 (i.e. progression free survival after both STZ based chemotherapy and Everolimus or the reverse order) as secondary endpoint. This information will be extremely valuable for the day to day clinical practice of pNETs oncologists

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of unresectable or metastatic, advanced pancreatic NET.
* Documented confirmation of pancreatic NET G1 or G2 as per European Neuroendocrine Society (ENETS) classification system.
* Patients from whom a paraffin-embedded primary tumour or metastasis block is available and to be sent by Courier.
* Before study inclusion, patients must show progressive disease documented by radiology 12 months prior to study inclusion. Treatment naive patients can be also included if the patient needs active treatment with either chemotherapy or everolimus.
* Presence of measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.0, documented by a Triphasic Computed Tomography (CT) scan or multiphase MRI radiological assessment.
* Previous treatment with somatostatin (SS) analogues is allowed. Only those patients with active functioning syndrome at entry can continue with SS analogues during the study.
* Adequate bone marrow and renal functions, and serum fasting cholesterol
* Women with child-bearing potential must have a negative serum pregnancy test.
* Written Informed Consent obtained according to local regulations

Exclusion Criteria:

* Previous treatment with chemotherapy and/or mTOR inhibitors or tyrosine kinase inhibitors.
* Immune therapy or radiation therapy within 4 weeks prior to the patient entering the study.
* Hepatic artery embolization within the last 6 months (1 month if there are other sites of measurable disease), or cryoablation/radiofrequency ablation of hepatic metastasis within 2 months of enrolment.
* Previous treatment with Peptide-Receptor Radionuclide Therapy (PRRT) within the last 6 months and/or without progression following PRRT.
* Uncontrolled diabetes mellitus.
* Any severe and/or uncontrolled medical conditions.
* Treatment with potent inhibitors or inducers of Cytochrome P450 3A4 (CYP3A) isoenzyme within 5 days immediately before the start of treatment.
* Patients on chronic treatment with corticosteroids or any other immunosuppressive agent.
* Patients known to be HIV seropositive.
* Known intolerance or hypersensitivity to everolimus or its excipients or other rapamycin analogues. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicinal product.
* Known intolerance or hypersensitivity to 5FU or STZ or its excipients (notice that this criterion includes patients with known deficit of dihydropyrimidine dehydrogenase deficiency -DPD).
* Pregnant, lactating women or fertile adults not using effective birth control methods.
* For administrative matters (insurance) patients ≥ 95 are not allowed during the trial.

Only those patients coming from the hospital pool will be included in SEQTOR trial (e.g. persons detained in an institution as a result of an official or court order are excluded).

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salazar Ramon, MD, PhD, Principal Investigator — Instituto Catalán de Oncologia, ICO-Hospitalet
Locations (37):
- Denmark (3):
  - Aarhus Aarhus University Hospital NET Centre (AUH-NET), Aarhus
  - Rigshospitalet NET CoE, University of Copenhagen, Copenhagen
  - Odense University Hospital, Odense
- France (8):
  - Brest Hopital Augustin Morvan, Institut de Cancero-Hemato, Brest, Brest Cedex
  - Clichy Neuroendocrine Tumor (NET) Center Hôpital Beaujon, Clichy, Clichy Cedex
  - Institut Gustave-Roussy, Villejuif, Paris
  - Hôpitaux Universitaires de Strasbourg Hôpital de Hautepierre, Strasbourg, Strasbourg Cedex
  - UTTIOM Unité Transversale de Thérapeutiques Innovantes en Oncologie Médicale CHU Angers, Angers
  - University Hospital of Bordeaux Hôpital Saint-André, Bordeaux
  - Hôpital Edouard Herriot, Lyon
  - Hôpital La Timone, Marseille
- Germany (10):
  - Bad Berka ChA Klinik für Innere Medizin, Bad Berka
  - Berlin Charité Universitätsmedizin, Berlin
  - Köln Universitätsklinikum Köln (AöR), Cologne
  - UKM Facharzt für Innere Medizin Gastroenterologie, Onkologische Gastroenterologie (DGVS), Halle
  - Medizinische Klinik und Poliklinik , Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Magdeburg Universitätsklinikum Magdeburg A. ö. R, Magdeburg
  - Mainz Universitätsmedizin, Mainz
  - Marburg Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - Interdisciplinary Center of Neuroendocrine Tumors of the GastroEnteroPancreatic System (GEPNET-KUM) at the University of Munich, München
  - Medizin II am Klinik und Poliklinik rechts der Isar, München
- Italy (2):
  - Istituto Nazionale Tumori (Fondazione G Pascale), Napoli, Naples
  - Istituto Europeo di Oncologia- IRCCS, Milan
- Netherlands (3):
  - Amsterdam Academic Medical Center, Amsterdam
  - UMCG / University of Groningen, Groningen
  - Maastricht UMC, Maastricht
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Instituto Catalán de Oncología de Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - HCU Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
- University Hospital, Uppsala, Sweden
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - The Royal Marsden, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No
As per GETNE guidelines and local laws

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A, Drug: Everolimus First: Everolimus (10mg/daily, oral) followed by STZ-5FU (injection/infusion; Moertel or Uppsala regime).
  Drug: Everolimus: 10mg/daily, oral. Number of Cycles: until progression or unacceptable toxicity develops.
  STZ-5FU: 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-5 every 6 weeks (Moertel) or 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-3, and then 1 day with 1g/m2 and 1 day 400mg/m2 5-FU every 3 weeks (Uppsala).
  Number of Cycles: until progression or unacceptable toxicity develops.
- Sequence B, Drug: STZ - 5FU First: STZ-5FU (injection/infusion; Moertel or Uppsala regime) followed by Everolimus (10 mg/ daily, oral)
  Drug: Everolimus: 10mg/daily, oral. Number of Cycles: until progression or unacceptable toxicity develops.
  STZ-5FU: 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-5 every 6 weeks (Moertel) or 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-3, and then 1 day with 1g/m2 and 1 day 400mg/m2 5-FU every 3 weeks (Uppsala).
  Number of Cycles: until progression or unacceptable toxicity develops.
Period: First Course Treatment
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Started | 72 | 69
Completed | 36 | 33
Not Completed | 36 | 36
Not completed — Adverse Event | 9 | 7
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Physician Decision | 9 | 9
Not completed — Death | 3 | 3
Not completed — Not reported reasons | 6 | 7
Not completed — Not treated | 3 | 3
Period: Second Course Treatment
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Started | 36 | 33
Completed | 36 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First | Total
Number analyzed (Participants) | 72 | 69 | 141
Age, Continuous [Median (Full Range); unit: years] | 58 [33 to 83] | 58 [33 to 80] | 58 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 41 | 44 | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Eastern cooperative oncology group (ECOG) performance status (PS) at baseline [Count of Participants; unit: Participants] — Baseline disease characteristics at inclusion to the study. ECOGis a scale that describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (death).
  Participants
    0 | 50 | 47 | 97
    1 | 20 | 22 | 42
    2 | 2 | 0 | 2
M-distant metastases at inclusion [Count of Participants; unit: Participants] — Presence of distant metastasis at the momento of randomization (baseline). Mx indicates that metastasis were assessed but the status of the patient regarding presence of metastasis could not be determined. M0 indicates no presence of distal metastasis. M1 indicates presence of distant metastasis and affectation of distant organs
  Participants
    Mx | 1 | 1 | 2
    M0 | 2 | 6 | 8
    M1 | 69 | 62 | 131
Location of metastases at randomization [Count of Participants; unit: Participants] — Number of patients who have distant organs affected by metastasis at randomization (Baseline). A patient may have more than one organ affected.
  Participants
    Bone | 7 | 10 | 17
    Lung | 2 | 3 | 5
    Liver | 61 | 56 | 117
    Lymph nodes | 4 | 6 | 10
Ki-67 [Count of Participants; unit: Participants] — Ki-67 is a protein found only in cells that are dividing. A high Ki-67 proliferation index means that many cells are dividing rapidly and that the cancer is likely to grow and spread.
  Here we used the categories used by the WHO classification for neuroendocrine tumors Population: patients with analyzable data
  Participants
    ≤ 2 | 9 | 14 | 23
    3-20 | 62 | 51 | 113
    Unknown | 1 | 4 | 5
Tumor Grade [Count of Participants; unit: Participants] — Tumor grade at randomization (baseline) using the World health organization (WHO) grading system for neuroendocrine tumors:
  G1: < 2 mitoses per 2 mm2 and/or Ki-67 index ≤ 2%, G2: 2-20 mitoses per 2 mm2 and/or Ki-67 index >2% and ≤ 20%
  Participants
    G1 | 9 | 12 | 21
    G2 | 63 | 55 | 118
    Unknown | 0 | 2 | 2
Number of previous systemic treatment lines [Count of Participants; unit: Participants]
  0 prior treatment lines | 36 | 43 | 79
  1 prior treatment line | 32 | 22 | 54
  2 prior treatment lines | 4 | 4 | 8
Previous treatments [Count of Participants; unit: Participants]
  Somatostatic analogs: Yes | 31 | 24 | 55
  Somatostatic analogs: No | 41 | 45 | 86
  Radiopharmaceuticals: Yes | 4 | 3 | 7
  Radiopharmaceuticals: No | 68 | 66 | 134
  Others: Yes | 1 | 1 | 2
  Others: No | 71 | 68 | 139

OUTCOME MEASURES:

1. Primary Outcome: First Progression Free Survival (PFS1)
Description: Proportion of patients who are alive without progression to Course 1 from the date of randomization in STZ based CT vs Everolimus arms
  Definitions for PFS rate for course 1 at 12 months:
  * No: number (proportion) of patients who were not alive and progression free according to the respective definition (main, conservative, and optimistic);
  * Yes: number (proportion) of patients who were alive and progression free according to the respective definition (main, conservative, and optimistic).
Time Frame: At 12 months
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs)
Measure: Number (95% Confidence Interval); unit: percentage of patients alive and PD-free
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 72 | 69
percentage of patients alive and PD-free | 71.4 [59.4 to 81.6] | 61.8 [49.2 to 73.3]
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.229, Regression, Cox; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.32 to 1.32]

2. Secondary Outcome: Second Progression Free Survival (Second PFS)
Description: PFS of Course 1 (PFS1) + interval between treatments + PFS of Course 2 (PFS2), where PFS1 represents progression free survival of Course 1 and PFS2 represents progression free survival of Course 2
Time Frame: Until the end of study every 12 weeks, approximately up to 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 72 | 69
months | 37.5 [27.1 to 53.7] | 32.6 [23.7 to 41.1]
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.135, Regression, Cox; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.90 to 2.19]

3. Secondary Outcome: Progression-free Survival (PFS) to First Treatment
Description: Time from the date of randomization to the date of first disease progression.
Time Frame: Throughout the study period every 12 weeks, approximately up to 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 72 | 69
months | 19.4 [16.8 to 27.6] | 22.7 [13.3 to 28.6]
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.474, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.77 to 1.75]

4. Secondary Outcome: Adverse Events (AEs) Rate
Description: Number of patients expiriencing adverse events, treatment-related AEs and serious adverse events (SAEs)
Time Frame: Throughout the study period in continous monitoring at every visit for approximately up to 5 years
Population: Patients who do not received study treatment were not included in the safety population to analyze safety.
  The outcome is reported per arm, as the trial was designed to report which sequential strategy is the best in overall. Most patients with panNETs progress and therefore will require to go through both treatments. The main scientific interest is the overall safety/efficacy.
Measure: Number; unit: Patients
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 69 | 66
Patients
  AEs | 68 | 62
  SAEs | 28 | 26
  Treatment-related AEs | 66 | 56

5. Secondary Outcome: Frequency of Dose Modifications to First Treatment
Description: Percentage of patients who require a dose reduction or interruption for management of adverse events during the study period
Time Frame: Throughout the study period, approximately up to 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving study treatment.
Measure: Number; unit: Patients
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 68 | 66
Patients | 41 | 9
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.001, Fisher Exact

6. Secondary Outcome: Best Overall Response (BOR) to First Study Treatment
Description: Best response achieved with the first study treatment according to RECIST V1.0
Time Frame: Throughout the study period, every 12 weeks up to approximately 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 69 | 66
Participants
  Complete response (CR) | 3 | 3
  Partial response (PR) | 5 | 17
  Stable disease (SD) | 58 | 35
  Progression of the disease (PD) | 2 | 9
  Not evaluable (NE) | 1 | 2

7. Secondary Outcome: Objective Response Rate (ORR) to First Study Treatment
Description: The ORR is defined as the number of patients having as their BOR to first treatment either Complete response (CR) or Partial Response (PR) measured by RECIST criteria version 1.0.
Time Frame: Throughout the study period every 12 weeks, up to approximately 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 69 | 66
Participants
  CR / PR | 8 | 20
  SD / PD / NE | 61 | 46
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.012, Fisher Exact

8. Secondary Outcome: Frequency of Dose Modifications to Second Treatment
Description: as for outcome 5
Time Frame: Throughout the study period, approximately up to 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving the second-line study treatment.
Measure: Number; unit: Patients
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 36 | 33
Patients | 5 | 18
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.001, Fisher Exact

9. Secondary Outcome: Overall Survival (OS)
Description: The median OS defined as the time from the date of randomization until death from any cause. This is estimated by kaplan meier method.
Time Frame: Throughout the study period, up to approximately 5 years
Population: Intention to treat population. The outcome is reported per arm rather than intervention, as the trial was designed to demonstrate which sequential strategy is the best in overall. Most patients with panNETs progress and therefore will require to go through both treatments. The main scientific interest is the overall safety/efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 72 | 69
months | 61.7 [49.1 to NA] — The interval have not reached | 50.6 [40.9 to 64.5]
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.168, Regression, Cox; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.86 to 2.37]

10. Secondary Outcome: Best Overall Response (BOR) to Second Study Treatment
Description: Best response achieved with the second study treatment according to RECIST V1.0
Time Frame: Throughout the study period, every 12 weeks up to approximately 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving the second treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 36 | 33
Participants
  Complete response (CR) | 1 | 0
  Partial response (PR) | 10 | 3
  Stable disease (SD) | 15 | 20
  Progression of the disease (PD) | 8 | 8
  Not evaluable (NE) | 2 | 2

11. Secondary Outcome: Objective Response Rate (ORR) to Second Study Treatment
Description: The ORR is defined as the number of patients having as their BOR to second treatment either Complete response (CR) or Partial Response (PR) measured by RECIST criteria version 1.0.
Time Frame: Throughout the study period every 12 weeks, up to approximately 5 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs) receiving second study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 36 | 33
Participants
  CR / PR | 11 | 3
  SD / PD / NE | 25 | 30
Statistical Analysis 1: Comparison: Sequence A, Drug: Everolimus First vs Sequence B, Drug: STZ - 5FU First; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.072, Fisher Exact

12. Other Pre Specified Outcome: Quality of Life Questionnaire (QLQ). The EORTC QLQ-C30 Global Health Status
Description: Patient self-reported quality of life (QoL) was assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire and the specific module for NETs, QLQ-GINET21.
  These questionnaires have a punctuation that ranges from 100 (best patient performance) to 0 (worse patient performance).
  Here we report the total QLQ-C30 score.
  Timepoints: Before any dose of study treatment (basal), before the first dose of the second treatment at line 2 cycle 1 (L2C1) and after completion of both treatments (EOT). Patients changed treatment line and ended both treatments after progression, therefore this outcome is not linked to specific reference timepoints but rather to a relevant disease stage which may happer early or latter in time. All assessments are performed obviously during trial duration, up to approximately 5 years.
Time Frame: Before any dose of study treatment (basal), before the first dose of the second treatment at line 2 cycle 1 (L2C1) and after completion of both treatments (EOT). See outcome measure description for further details.
Population: Patients completing the QLQ questionnaires at any timepoint.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Sequence A, Drug: Everolimus First | Sequence B, Drug: STZ - 5FU First
Number analyzed (Participants) | 47 | 49
Score
  Basal | 78.3 (17.6) | 77.8 (12.1)
  L2C1: number analyzed (Participants) | 18 | 20
  L2C1 | 75.1 (16) | 84.1 (9.5)
  EOT: number analyzed (Participants) | 20 | 13
  EOT | 68.4 (15.2) | 75.4 (17.9)

13. Secondary Outcome: Progression-free Survival (PFS) to Second Treatment
Description: Time from the date of first dose of second treatment to the date of second disease progression.
Time Frame: Throughout the study period every 12 weeks, approximately up to 2 years
Population: Patients diagnosed advanced progressive pancreatic neuroendocrine tumours (pNETs)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sequence A, Drug: STZ-5FU Second: STZ-5FU: 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-5 every 6 weeks (Moertel) or 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-3, and then 1 day with 1g/m2 and 1 day 400mg/m2 5-FU every 3 weeks (Uppsala).
  Number of Cycles: until progression or unacceptable toxicity develops.
- Sequence B, Drug: Everolimus Second: STZ-5FU (injection/infusion; Moertel or Uppsala regime) followed by Everolimus (10 mg/ daily, oral)
  Drug: Everolimus: 10mg/daily, oral. Number of Cycles: until progression or unacceptable toxicity develops.
Arm/Group | Sequence A, Drug: STZ-5FU Second | Sequence B, Drug: Everolimus Second
Number analyzed (Participants) | 36 | 33
months | 8.8 [5.2 to 30.2] | 9.5 [6.6 to 19.3]
Statistical Analysis 1: Comparison: Sequence A, Drug: STZ-5FU Second vs Sequence B, Drug: Everolimus Second; significant differences between both arms is assumed in case p-val < 0.05; Test type: Superiority; p = 0.079, Log Rank; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [0.94 to 2.73]

ADVERSE EVENTS:
Time Frame: From the time the patient signs IC for the study until 30 days after the intake of the last dose of treatment; up to approximately 5 years
Description: Adverse events and deaths reported "per intervention" (e.g., "Everolimus" and "STZ-5FU") as pre-specified in the protocol.
Groups:
- Everolimus: Drug: Everolimus: 10mg/daily, oral. Number of Cycles: until progression or unacceptable toxicity develops.
- STZ - 5FU: STZ-5FU: 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-5 every 6 weeks (Moertel) or 0,5g/m2 STZ on days 1-5 and 400mg/m2 5-FU on days 1-3, and then 1 day with 1g/m2 and 1 day 400mg/m2 5-FU every 3 weeks (Uppsala).
  Number of Cycles: until progression or unacceptable toxicity develops.
Arm/Group | Everolimus | STZ - 5FU
All-Cause Mortality (participants affected / at risk) | 26/105 | 35/104
Serious Adverse Events (participants affected / at risk) | 28/105 | 26/104
Other Adverse Events (participants affected / at risk) | 68/105 | 62/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=105) | STZ - 5FU (N=104)
Fever (General disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Sepsis (Infections and infestations) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Malaise (General disorders) | 2 | 0
Infection without focus (Infections and infestations) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine increased (Investigations) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Localized edema (Skin and subcutaneous tissue disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Acute cholangitis (Hepatobiliary disorders) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Increased urea (Investigations) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Renal Calculi (Renal and urinary disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Urotelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liver metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Renal and urinary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=105) | STZ - 5FU (N=104)
Fever (General disorders) | 14 | 5
Abdominal pain (Gastrointestinal disorders) | 14 | 17
Hyperglycemia (Metabolism and nutrition disorders) | 23 | 9
Constipation (Gastrointestinal disorders) | 10 | 15
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 | 0
Fatigue (General disorders) | 39 | 37
Nausea (Gastrointestinal disorders) | 21 | 26
Urinary tract infection (Infections and infestations) | 11 | 3
Anemia (Blood and lymphatic system disorders) | 10 | 3
Weight loss (Investigations) | 9 | 5
Lung infection (Infections and infestations) | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Creatinine increased (Investigations) | 4 | 6
Non-cardiac chest pain (General disorders) | 4 | 4
Mucositis oral (Gastrointestinal disorders) | 34 | 16
Diarrhea (Gastrointestinal disorders) | 26 | 19
Rash acneiform (Skin and subcutaneous tissue disorders) | 26 | 4
Edema limbs (General disorders) | 17 | 5
Anorexia (Metabolism and nutrition disorders) | 16 | 12
Vomiting (Gastrointestinal disorders) | 12 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 3
Platelet count decreased (Blood and lymphatic system disorders) | 10 | 7
Flu like symptoms (General disorders) | 10 | 9
Cholesterol high (Investigations) | 10 | 2
Alanine aminotransferase increased (Investigations) | 8 | 2
Dysgeusia (Nervous system disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Hypertension (Vascular disorders) | 8 | 1
Headache (Nervous system disorders) | 7 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Proteinuria (Renal and urinary disorders) | 6 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 1
Stomach pain (Gastrointestinal disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Mouth ulcer (Gastrointestinal disorders) | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 4 | 2
GGT increased (Investigations) | 4 | 0
Upper respiratory infection (Infections and infestations) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 8
Nail ridging (Skin and subcutaneous tissue disorders) | 4 | 0
Pharyngitis (Infections and infestations) | 4 | 0
Skin infection (Infections and infestations) | 4 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 5
Thromboembolic event (Vascular disorders) | 2 | 4
Pain in extremity (General disorders) | 3 | 6
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Cramps (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 1 | 4
Alkaline phosphatase increased (Investigations) | 3 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT02246127/Prot_SAP_000.pdf